CLINICAL TRIAL: NCT06830395
Title: A Phase II Clinical Study to Evaluate the Safety and Efficacy of CM313 (SC) Injection in Subjects With Primary IgA Nephropathy
Brief Title: Study of CM313 in Subject With IgA Nephropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM313-105101
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part A: CM313 low dose (Experimental)
  Interventions: Biological: CM313
- Part A: CM313 high dose (Experimental)
  Interventions: Biological: CM313
- Part B: CM313 low dose with low frequency (Experimental)
  Interventions: Biological: CM313
- Part B: CM313 low dose with high frequency (Experimental)
  Interventions: Biological: CM313
- Part B: Placebo matching the volume of low dose CM313 (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B: CM313 high dose with low frequency (Experimental)
  Interventions: Biological: CM313
- Part B: CM313 high dose with high frequency (Experimental)
  Interventions: Biological: CM313
- Part B: Placebo matching the volume of high dose CM313 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM313 — CM313(SC) injection
  Arms: Part A: CM313 high dose; Part A: CM313 low dose; Part B: CM313 high dose with high frequency; Part B: CM313 high dose with low frequency; Part B: CM313 low dose with high frequency; Part B: CM313 low dose with low frequency
Drug: Placebo — Matched placebo
  Arms: Part B: Placebo matching the volume of high dose CM313; Part B: Placebo matching the volume of low dose CM313

SUMMARY:
This study is divided into two parts (Part A and Part B). This study aims to evaluate the safety and efficacy of CM313 in subjects with primary Immunoglobulin A nephropathy(IgAN), while also observing its Pharmacokinetics(PK) characteristics, Pharmacokinetics(PD) effects, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend the research study and voluntarily signing the informed consent form (ICF).
* Renal biopsy report supporting diagnosis of primary IgAN within 8 years prior to the screening visit.
* Estimated Glomerular Filtration Rate (eGFR) (using the Chronic Kidney Disease Epidemiology Collaboration formula) ≥ 30 mL/min/1.73 (m*m) at screening and baseline.
* Prior to the baseline visit, all subjects must have received standard care treatment, including good blood pressure control and a stable treatment of a maximum recommended or maximum tolerated dose of angiotensin-converting enzyme inhibitors(ACEI) or Angiotensin receptor blocker(ARB) for at least 12 weeks.
* 24-hour urinary protein-to-creatinine ratio (24h-UPCR) ≥ 0.75 g/g or 24-hour urinary protein excretion (24h-UPE) ≥ 1 g/d during the screening and baseline periods.

Exclusion Criteria:

* Secondary IgAN judged by the investigator: Secondary IgAN may be associated with Henoch-Schonlein purpura, hepatic cirrhosis, coeliac disease, human immunodeficiency virus (HIV) infection, dermatitis herpetiformis, seronegative arthritis, small cell carcinoma, lymphoma, disseminated tuberculosis, obliterative bronchiolitis, inflammatory bowel disease, familial Mediterranean fever, etc.
* Known allergy to monoclonal antibody drugs or to the excipients of CM313.
* Presence of rapidly progressive glomerulonephritis (RPGN), defined as 50% decline in eGFR within 3 months prior to randomization and/or crescent formation in more than 50% of glomeruli in a renal pathological specimen.
* Confirmed acute kidney injury (AKI) within 4 weeks prior to randomization.
* Vaccination of any live vaccine within 30 days prior to dosing or planned vaccination during the study period.
* History of transplantation (any solid organ transplant, including renal transplant, bone marrow transplant, etc.) or plan to undergo renal transplantation during the study.
* History of severe recurrent or chronic infection.
* Malignant tumor within 5 years prior to screening (except for completely cured cervix carcinoma in situ and non-skin squamous cell carcinoma metastatic or basal cell carcinoma).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to 108 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Jicheng Lv, Principal Investigator — Peking University Frist Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China